CLINICAL TRIAL: NCT03981770
Title: Characterisation of Gut Microbiota, Bispectral Index Data and Plasma Kynurenine in Patients Undergoing Thyroid Surgery
Status: Completed | Type: Observational
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Wen-fei Tan, Professor, China Medical University, China
Other Study IDs: 20190607
Record Dates: First submitted 2019-06-07; First posted 2019-06-11 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Sleep Deprivation
MeSH Terms: conditions — Sleep Deprivation | interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group good sleepers: Duration of sleep was defined as the duration of all Bispectral Index data below 80 in the 12 hours of monitoring (from 18:00pm to 06:00am). Sleeping time are more than four hours.
  Interventions: Drug: General anesthesia
- Group poor sleepers: Duration of sleep was defined as the duration of all Bispectral Index data below 80 in the 12 hours of monitoring (from 18:00pm to 06:00am). Sleeping time are less than four hours.
  Interventions: Drug: General anesthesia

INTERVENTIONS:
Drug: General anesthesia — For maintenance of propofol anesthesia, total intravenous anesthesia was administered by using propofol (Fresenius Kabi, Austria GmbH) at a plasma target concentration (Marsh pharmacokinetic model software) of 2.5-4 μg/ml. Remifentanil (0.2-0.5 μg/kg/min) was given to all patients during the operation.

SUMMARY:
The study is a case-controlled observational trial. Forty patients will be divided into 2 groups (good or poor sleepers) depending on their first postoperative night Bispectral index data. Firstly, this study aims to characterise the lung microbiota in patients treated with thyroid surgery. Secondly, it aims to evaluate microbiota and its influence on plasma kynurenine.

DETAILED DESCRIPTION:
The study is a case-controlled observational trial. Forty patients will be divided into 2 groups (good or poor sleepers) depending on their first postoperative night Bispectral index data. Firstly, this study aims to characterise the lung microbiota in patients treated with thyroid surgery. Secondly, it aims to evaluate microbiota and its influence on plasma kynurenine.

ELIGIBILITY:
Inclusion Criteria:

* ethnic Chinese;
* age, 18 to 65 years old;
* American Society of Anaesthesiologists (ASA) physical status I or II

Exclusion Criteria:

* Cognitive difficulties
* Affiliated with the Social Security System
* Partial or complete gastrectomy
* Previous esophageal surgery
* Inability to conform to the study's requirements
* Deprivation of a right to decide by an administrative or juridical entity
* Ongoing participation or participation in another study <1 month ago

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male
Study Population: The study is a case-controlled observational trial. Forty patients will be divided into 2 groups (good or poor sleepers) depending on their first postoperative night Bispectral index data. Firstly, this study aims to characterise the lung microbiota in patients treated with thyroid surgery. Secondly, it aims to evaluate microbiota and its influence on plasma kynurenine.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
gut microbiota | the first postoperative night
  this study will characterise the gut microbiota in 2 groups of 30 patients.

SECONDARY OUTCOMES:
Bispectral index data | the first postoperative night
  this study will characterise the Bispectral index data in 2 groups of 30 patients
plasma kynurenine concentrations | baseline and the first postoperative night
  this study will characterise the plasma kynurenine concentrations in 2 groups of 30 patients

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No